CLINICAL TRIAL: NCT03468738
Title: Investigation of the Transfusion Practices in Surgical Patients in Turkey
Acronym: CeKATU
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Collaborators: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Associate Professor, Diskapi Teaching and Research Hospital
Other Study IDs: Dilek Yazıcıoglu Unal
Record Dates: First submitted 2018-03-11; First posted 2018-03-19 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Surgery; Blood Loss, Surgical; Blood Loss Anemia; Blood Transfusion; Anemia; Coagulation Disorder
MeSH Terms: conditions — Blood Loss, Surgical; Anemia; Hemostatic Disorders | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood transfusion — Transfusion of blood products in the perioperative period in patients undergoing major surgery

SUMMARY:
The aim of this study is to describe the transfusion practices in patients undergoing major surgery in Turkey. The transfusion rates of red blood cells (RBC), fresh frozen plasma (FFP) and platelets; the transfusion predictors and transfusion related patient outcomes are investigated.

DETAILED DESCRIPTION:
Patient Blood Management (PBM) is an evidence based multidisciplinary approach for the care of patients who may need blood transfusion. The aim of PBM is achieving better patient outcomes by focusing on the patients' own blood as a source.

To date PBM is considered "good transfusion practice" and is being implemented in a growing number of countries. The Turkish Society of Anesthesiologists PBM Task Force is working on this subject since 4 years and decided to conduct a study. Before starting a PBM program, the transfusion practices of clinicians working at diverse surgical fields; differences between current transfusion practices and PBM strategies; the areas for improvement and the obstacles that could prevent change could be identified with this study. Data collection will also serve to identify the current situation as a reference and to control the achievement of the PBM's aim: improving clinical outcomes. These data will be refered as The Turkish National Perioperative Transfusion Study (TULIP TS) data.

The aim of this study is to describe the transfusion practices in patients undergoing major surgery in Turkey.

The study evaluates i. The perioperative transfusion rates of RBCs, FFP and platelets. ii. With which reasons the anesthesiologists decide to transfuse a patient (co morbidities of the patients, physiologic transfusion triggers, hemoglobin trigger, uncontrolled bleeding, on request from surgeon etc.).

iii. The relation of transfusion and the patients co-morbidity index, the P POSSUM score and SORT score; anesthesia methods; monitorisation methods (hemodynamic, coagulation); amount of bleeding; type of surgery; type of hospital.

iv. The relation of transfusion and patient outcomes (unanticipated ICU admission, prolonged ICU stay, acute renal failure, thromboembolic events, ischemic events, pulmonary complications, cardiac advers events, infections, acute respiratory distress, infection, all-cause mortality).

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing major elective surgery

Exclusion Criteria:

Trauma patients, emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing major elective surgery in General surgery Orthopedics Urology Transplantation surgery Neurosurgery Gynecology and obstetrics Cardiovascular surgery
Sampling Method: Probability Sample
Enrollment: 6481 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Preoperative amount of blood products transfused | Before surgery at day 0
  Preoperative amount of blood products: RBCs,FFP and platelets transfused
Intraoperative amount of blood products transfused | During surgery at day 0
  Intraoperative amount of blood products: RBC's,FFP and platelets transfused
Postoperative amount of blood products transfused | 24 hours after surgery
  Postoperative amount of blood products: RBCs,FFP and platelets transfused

SECONDARY OUTCOMES:
Preoperative transfusion indications | Before surgery at day 0
  The reasons to decide to transfuse (factors determining transfusion) blood products
Intraoperative transfusion indications | During surgery at day 1
  The reasons to decide to transfuse (factors determining transfusion) blood products
Postoperative transfusion indications | 24 hours after surgery
  The reasons to decide to transfuse (factors determining transfusion) blood products
Unanticipated ICU admission | After surgery at day 1
  Whether the patient had an unanticipated ICU admission
Prolonged length of stay in ICU | After surgery at day 2
  Whether the patient had a prolonged length of stay in ICU
Acute renal failure | After surgery at day 2
  Whether the patient had acute renal failure
Thromboembolic event | After surgery at day 2
  Whether the patient had a thromboembolic event concerning lungs (pulmonary embolism), brain (stroke), gastrointestinal tract, kidneys, or extremities etc.
Ischemic event | After surgery at day 2
  Whether the patient had an ischemic event concerning heart, nervous system,limb, gastrointestinal tract etc.
Infection | After surgery at day 2
  Whether the patient had infection: wound, pneumonia, urinary, sepsis etc.
Acute respiratory distress | After surgery at day 2
  Whether the patient had acute respiratory distress
Mortality | after surgery at day 30
  Whether the patient died: all cause mortality
Preoperative anemia | Before surgery at day 0
  Whether the patient had anemia (Hemoglobin male < 13 female < 12 g/dL)
Preoperative coagulopathy | Before surgery at day 0
  Whether the patient had coagulopathy due to disease or drugs
Pretransfusion hemoglobin values | Before surgery at day 0
  The hemoglobin concentration before transfusion
Pretransfusion hemoglobin values | During surgery at day 1
  The hemoglobin concentration before transfusion
Pretransfusion hemoglobin values | After surgery at day 2
  The hemoglobin concentration before transfusion
Advers cardiac events | After surgery at day 30
  Whether the patient had an advers cardiac event: myocardial infaction; non fatal cardiac arest; arrhytmia; cardiogenic pulmonary edema etc

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Unal, Assoc Prof, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (61):
- Turkey (Türkiye) (61):
  - Acibadem University Mehmet Ali Aydinlar Atakent Hospital, Ankara
  - Ankara University Cebeci Medical Center, Ankara
  - Ankara University Ibni Sina Hospital, Ankara
  - Başkent University Ankara Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Private Cankaya Hospital, Ankara
  - Ufuk University Medical Faculty Dr. Ridvan Ege Training and Research Hospital, Ankara
  - University of Health sciences Ankara Child Health and Diseases Hematology Oncology Training and research Hospital, Ankara
  - University of Health Sciences Ankara Numune Training and Research Hospital, Ankara
  - University of Health Sciences Ankara Training and Research Hospital, Ankara
  - University of Health Sciences Diskapi Yildirim Beyazit Trainig Research Hospital, Ankara
  - University of Health Sciences Dr Abdurrahman Yurtaslanı Ankara Oncology Training and Research Hospital, Ankara
  - University of Health Sciences Kecioren Training and Research Hospital, Ankara
  - University of Health Sciences Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara
  - University of Health Sciences Yenimahalle Training and Research Hospital, Ankara
  - University of Health Sciences Zubeyde Hanim Gynecology and Maternity Training and Research Hospital, Ankara
  - University of Technology and Economics Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - University of Health Sciences Antalya Training and Research Hospital, Antalya
  - Balikesir University Training and Research Hospital, Balıkesir
  - Uludağ University Medical Faculty, Bursa
  - University of Health Sciences Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Hitit University Corum Erol Olcok Training and Research Hospital, Çorum
  - Trakya University Medical Faculty, Edirne
  - Fırat University Medical Faculty, Elâzığ
  - Erzincan University Mengucek Gazi Training and Research Hospital, Erzincan
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir
  - Suleyman Demirel University Medical Faculty, Isparta
  - Acibadem University Altunizade Hospital, Istanbul
  - Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul
  - Istanbul University Medical Faculty, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - University of Health Sciences Fatih Sultan Mehmet Training and Research Hospital, Istanbul
  - University of Health Sciences Haydarpasa Numne Training and Research Hospital, Istanbul
  - University of Health Sciences Istanbul Training and Research Hospital, Istanbul
  - University of Health Sciences Kanuni Sultan Suleyman Training and Research Hospital, Istanbul
  - University of Health Sciences Okmeydanı Training and Research Hospital, Istanbul
  - University of Health Sciences Umraniye Training and Research Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - University of Health Sciences Bozyaka Training Research Hospital, Izmir
  - University of Health Sciences İzmir Tepecik Training and Research Hospital, Izmir
  - Sutcu Imam University Medical Faculty, Kahramanmaraş
  - Erciyes University Medical Faculty, Kayseri
  - University of Health Sciences Kayseri Training and Research Hospital, Kayseri
  - Anadolu Health Center Hospital, Kocaeli
  - University of Health Sciences Derince Training and Research Hospital, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty Center for Health and Research, Konya
  - Selcuk University Medical Faculty, Konya
  - University of Health Sciences Konya Training and Research Hospital, Konya
  - Inonu University Liver Transplantation Institute, Malatya
  - Manisa Celal Bayar University Medical Faculty Hafsa Sultan Hospital, Manisa
  - Mersin University Medical Faculty, Mersin
  - Ordu University Medical Faculty, Ordu
  - Osmaniye State Hospital, Osmaniye
  - Ondokuz Mayıs University Medical Faculty, Samsun
  - Namık Kemal University Medical Faculty, Tekirdağ
  - Karadeniz Technical University Medical Faculty Farabi Hospital, Trabzon
  - Tunceli State Hospital, Tunceli
  - Van Yuzuncuyıl University Medical Faculty Dursun Odabası Center, Van
  - Bulent Ecevit University Medical Faculty Center for Health and Research, Zonguldak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotze A, Carter LA, Scally AJ. Effect of a patient blood management programme on preoperative anaemia, transfusion rate, and outcome after primary hip or knee arthroplasty: a quality improvement cycle. Br J Anaesth. 2012 Jun;108(6):943-52. doi: 10.1093/bja/aes135. PMID 22593128
- [Background] Meier J, Filipescu D, Kozek-Langenecker S, Llau Pitarch J, Mallett S, Martus P, Matot I; ETPOS collaborators. Intraoperative transfusion practices in Europe. Br J Anaesth. 2016 Feb;116(2):255-61. doi: 10.1093/bja/aev456. PMID 26787795
- [Background] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234
- [Background] Kalil AC, Mattei J, Florescu DF, Sun J, Kalil RS. Recommendations for the assessment and reporting of multivariable logistic regression in transplantation literature. Am J Transplant. 2010 Jul;10(7):1686-94. doi: 10.1111/j.1600-6143.2010.03141.x. PMID 20642690